CLINICAL TRIAL: NCT04788628
Title: Effects of Auditory Stimulation on Coordinated Non-REM Sleep Oscillations and Memory in Epilepsy Inpatients With Implanted Hippocampal Electrodes
Brief Title: Auditory Stimulation Effects on Sleep and Memory in Patients With Epilepsy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Dara S. Manoach, PhD, Professor, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2020P003959
Record Dates: First submitted 2021-02-25; First posted 2021-03-09 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Epilepsy
Keywords: Sleep; Memory; Auditory stimulation; Spindles; Intracranial monitoring; Hippocampal ripples; Slow oscillations
MeSH Terms: conditions — Epilepsy | interventions — BaseLine dental cement; Acoustic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Epilepsy inpatients (Experimental): Epilepsy inpatients with implanted hippocampal electrodes and continuous scalp EEG monitoring
  Interventions: Other: Baseline; Other: Motor procedural memory task; Other: Motor procedural memory task plus auditory stimulation

INTERVENTIONS:
Other: Baseline — Hippocampal and scalp EEG monitoring during overnight sleep
Other: Motor procedural memory task — Training on the finger tapping MST prior to monitored overnight sleep with MST testing the following morning
Other: Motor procedural memory task plus auditory stimulation — Training on the finger tapping MST prior to monitored overnight sleep that includes auditory stimulation, with MST testing the following morning

SUMMARY:
This study will investigate the role of coordinated brain rhythms during sleep in memory consolidation and determine whether playing precisely timed brief bursts of noise can enhance these rhythms and improve memory in epilepsy inpatients with implanted hippocampal electrodes.

DETAILED DESCRIPTION:
The investigators will test the hypotheses that coordinated brain rhythms during nonrapid eye movement sleep are associated with memory consolidation and can be enhanced with auditory stimulation (playing precisely timed brief bursts of quiet noise) to improve memory. The investigators will measure differences in sleep and memory performance in epilepsy inpatients with implanted hippocampal electrodes and continuous full scalp EEG monitoring under three overnight sleep conditions: a baseline night; a memory night during which sleep-dependent memory consolidation is assessed with the finger tapping motor sequence task (MST) with training prior to sleep and testing the next morning; and a stimulation night during which participants train on the MST, have precisely timed auditory stimulation during the sleep that follows, and are tested on the MST in the morning.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients with epilepsy
* Aged 12-65
* Undergoing clinically indicated continuous scalp and intracranial EEG monitoring with implanted hippocampal electrodes
* Fluent in English
* Able to give informed consent/assent (for minors aged 12-17 or adults with an appointed guardian)

Exclusion Criteria:

* Intellectual disability impairing ability to perform task
* Motor problems that preclude finger tapping task
* Previous surgery anticipated to disrupt coordination of sleep oscillations in the circuitry of interest

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-01-21 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Changes in slow oscillation-spindle-hippocampal ripple coupling | Three nights of sleep within three weeks
  Changes in the coupling of slow oscillations with spindles and hippocampal ripples during non-Rapid Eye Movement (NREM) sleep as measured by scalp and intracranial EEG between baseline, memory, and auditory stimulation nights.

SECONDARY OUTCOMES:
Changes in sleep-dependent consolidation of motor procedural memory | Three nights of sleep within three weeks
  Changes in sleep-dependent improvement of motor procedural memory performance on the finger tapping motor sequence task (MST) between baseline, memory, and auditory stimulation nights. Different sequences are employed for the memory and auditory stimulation nights in a counter-balanced order.
Changes in slow oscillations | Three nights of sleep within three weeks
  Changes in slow oscillations during non-rapid eye movement (NREM) sleep as measured by EEG between the baseline, memory, and auditory stimulation nights
Changes in sleep spindles | Three nights of sleep within three weeks
  Changes in sleep spindles during non-rapid eye movement (NREM) sleep as measured by EEG between baseline, memory, and auditory stimulation nights
Changes in hippocampal ripples | Three nights of sleep within three weeks
  Changes in hippocampal ripples during non-rapid eye movement (NREM) sleep as measured by intracranial EEG between baseline, memory, and auditory stimulation nights

CONTACTS AND LOCATIONS:
Overall Officials: Dara Manoach, PhD, Principal Investigator — Professor
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The PI will disseminate results through presentations at public lectures, scientific institutions and meetings, and/or publications in major journals. The institution and the PI will adhere to the NIH Grants Policy on Sharing of Unique Research Resources including the Sharing of Biomedical Research Resources. Prevailing standards and guidelines in documenting and depositing data sets will be followed. Specifically, quality-controlled data used in publications will be deidentified and made available to requesting scientists, starting one year following the completion of the project. Workflows will be documented and will allow any external groups to reproduce results from the raw data. The PI will be responsible for overseeing the sharing the data. Raw and summary data will be submitted to the appropriate NIMH Data Archive annually, including The National Database for Clinical Trials Related to Mental Illness (NDCT).
Time Frame: Data will be available one year following the completion of the project.